CLINICAL TRIAL: NCT05273983
Title: Pilot Study of a Brief Behavioural Activation Intervention for Depressed Patients in Primary Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator medical leave
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS25208
Record Dates: First submitted 2022-02-01; First posted 2022-03-10 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Major Depressive Disorder
Keywords: Behavioural activation; Psychological treatment; Primary care
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioural Activation Treatment (Experimental): Two intervention sessions with a psychologist and an use of a mobile scheduling app over the course of 6 weeks.
  Interventions: Behavioral: Behavioural Activation

INTERVENTIONS:
Behavioral: Behavioural Activation — The intervention will span 6 weeks, including two intervention sessions with the primary care psychologist, and 6-weeks use of a mobile activity scheduling app (Strides). In the first intervention session, the psychologist would provide psychoeducation about depression, therapeutic rationale of behavioural activation, aid the patient in identifying their values and corresponding activities that may correspond with their values, introduce the mobile app, and help the patient schedule initial activities/goals. The second intervention session, which would be flexibly scheduled according to patient need, would focus on troubleshooting/clarification of previously discussed topics.

SUMMARY:
This study will explore the effectiveness of a brief psychological intervention for depressed outpatients in primary care. Participants will attend two intervention sessions with a psychologist and use a mobile activity/goal setting application for 6 weeks.

DETAILED DESCRIPTION:
This study will evaluate the feasibility and effectiveness of a two-session psychologist-led behavioural activation intervention, with adjunctive use of a free activity/goal setting app, for depressed patients in primary care. Outpatients in primary care with Major Depressive Disorder will be recruited to complete two intervention sessions with the primary care psychologist, as well as use the mobile activity scheduling app for 6 weeks. Symptom measures will be administered prior to both intervention sessions and 6-weeks after the first intervention session.

ELIGIBILITY:
Inclusion Criteria:

* Depression is the primary concern;
* Score of 10 or greater on a depression screening tool;
* Have access to an iPhone or iPad.

Exclusion Criteria:

* Another psychological disorder is the primary concern (e.g., anxiety disorder, personality disorder);
* Concurrent alcohol or drug use disorder;
* Unstable dose of psychotropic medication (i.e., any psychotropic medication doses will need to be stable for at least four weeks prior to enrolment);
* Current participation in other regular psychological treatment (e.g., cognitive behavioral therapy, counselling);
* At a high risk/emergent risk for suicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Change in depression symptoms as measured by the Patient Health Questionnaire-9 item (PHQ-9) | Change in score from baseline to 3 weeks
  This survey will be completed online. Participants will answer 9-items assessing symptoms and severity of depression, on a four-option scale from 0 (not at all) to 3 (nearly every day). A sum of the items produces a Total Score from 0 to 27. Higher scores indicate greater depression symptomology.
Change in depression symptoms as measured by the Patient Health Questionnaire-9 item (PHQ-9) | Change in score from baseline to 6 weeks.
  This survey will be completed online. Participants will answer 9-items assessing symptoms and severity of depression, on a four-option scale from 0 (not at all) to 3 (nearly every day). A sum of the items produces a Total Score from 0 to 27. Higher scores indicate greater depression symptomology.

SECONDARY OUTCOMES:
Change in anxiety symptoms as measured by the Generalized Anxiety Disorder-7 item Scale (GAD-7) | Change in score from baseline to 6 weeks
  This survey will be completed online. Participants will answer 7-items assessing symptoms and severity of generalized anxiety, on a four-option scale from 0 (not at all) to 3 (nearly every day). A sum of the items produces a Total Score form 0 to 21. Higher scores indicate greater anxiety symptomology.
Change in perceived life impairment as measured by the Work and Social Adjustment Scale (WSAS) | Change in score from baseline to 3 weeks
  This survey will be completed online. Participants will answer 5-items assessing perceived impairment in important life domains due to their depression, on a eight-option scale from 0 (no impairment at all) to 8 (very severe impairment). A sum of the items produces a Total Score from 0 to 40. Higher scores indicate greater perceived impairment.
Change in perceived life impairment as measured by the Work and Social Adjustment Scale (WSAS) | Change in score from baseline to 6 weeks
  This survey will be completed online. Participants will answer 5-items assessing perceived impairment in important life domains due to their depression, on a eight-option scale from 0 (no impairment at all) to 8 (very severe impairment). A sum of the items produces a Total Score from 0 to 40. Higher scores indicate greater perceived impairment.

OTHER OUTCOMES:
Treatment credibility and expectancy as measured by the Treatment Credibility and Expectancy Questionnaire (CEQ) | Baseline
  This survey will be completed online. Participants will answer six-items assessing their expectancy and credibility regarding the treatment, on a nine-option scale. A sum of the items produces a Total Score from 6 to 54. Higher scores indicate greater expectancy/credibility regarding the treatment and possible outcomes.
Quality of service as measured by the Client Satisfaction Questionnaire (CSQ-8) | The CSQ-8 will be completed six-weeks after baseline
  This survey will be completed online. Participants will answer eight-items assessing participant satisfaction with their treatment experience, on a four-option scale. A sum of the items produces a Total Score from 8 to 32. Higher scores indicate greater participant satisfaction.
Mobile app engagement as measured by an engagement questionnaire. | The engagement questionnaire will be completed six-weeks after baseline..
  This survey will be completed online. Participants will answer two-items assessing how often they used the mobile app over the six-weeks and how many activities they scheduled a week on average, through multiple choice options. Higher frequency of usage will indicate higher levels of engagement or treatment adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hebert, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Deer Lodge Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Result] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Result] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Result] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370